CLINICAL TRIAL: NCT03190408
Title: Observation of Variation in Fluids Administered and Characterization of Vasopressor Requirements in Shock
Brief Title: Variation in Fluids Administered in Shock
Acronym: VOLUME
Status: Completed | Type: Observational
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-7860
Record Dates: First submitted 2017-06-14; First posted 2017-06-16 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Shock
MeSH Terms: conditions — Shock | interventions — Fluid Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Shock
  Interventions: Other: Fluids

INTERVENTIONS:
Other: Fluids — Fluids Administered in Shock

SUMMARY:
To conduct a multicenter observational cohort study to determine the variability in fluid resuscitation in shock in a broad range of areas in hospitals and treatment areas.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years admitted to the participating hospital.
* Patients in the emergency department, intensive care unit, PACU, or any hospital floor. For patients not in the ICU, there must be plans to transfer to an intensive care unit when an ICU bed is available for patient.
* Patients with shock as defined by:
* Need for vasopressor (dopamine, norepinephrine, or epinephrine at any dose) to keep MAP > 65 mmHg Or
* Systolic BP < 90 mmHg

Exclusion Criteria:

* Patients previously enrolled into this study.
* Patients who were in the operating room at time of shock and fluid bolus.
* Patients admitted to an ICU after cardiac surgery Patients with primarily cardiogenic shock as etiology for their shock
* Patients transferred from another hospital or emergency room to the study hospital.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with shock
Sampling Method: Non-Probability Sample
Enrollment: 1639 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Method used to guide volume resuscitation | 7 days
  Characterize the method used to guide volume resuscitation and vasopressor use in patients with shock

CONTACTS AND LOCATIONS:
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States